CLINICAL TRIAL: NCT04184076
Title: Randomized Controlled Trial of Time-Restricted Feeding (TRF) in Acute Ischemic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201903100RINA
Record Dates: First submitted 2019-11-17; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-07

CONDITIONS: Fasting
Keywords: fasting; safety; compliance; ischemic stroke; time restricted feeding
MeSH Terms: conditions — Fasting; Patient Compliance; Ischemic Stroke; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary counseling alone (No Intervention): 1. Controls will be instructed to maintain their weight throughout the trial, and not to change their eating or physical activity habits. Controls will visit the research center on a weekly basis for weigh-ins. Body composition and metabolic disease risk variables will be assessed in control subjects every 12 weeks.
  2. Subjects will complete a 3-d food record (2 regular day and 1 holiday) each week during the experiment.
  3. The blood draws will be taken at approximately 11:00 am. The following analyzes will be measured in plasma samples: ketones, fasting glucose, fasting insulin, hemoglobin A1c, liver function, renal function, albumin, lipid profiles, MMP-9, IL-6, TNF-alpha, exosome markers (phospho-IRS1, phospho-Tau, Abeta1-42). Metabolomic and lipidomic analyses will be performed on the baseline and 3-month time point plasma samples.
- Time-restricted feeding (TRF) with dietary counseling (Experimental): 1. Subjects will be instructed to eat ad libitum from 10:00 to 18:00 h daily, and fast from 18:00 to 10:00 h daily. During the 8-h feeding window, there will be no restrictions on types or quantities of foods consumed. During the fasting period, subjects will be encouraged to drink plenty of water and will be permitted to consume energy-free beverages.
  2. Subjects will complete a 3-d food record (2 regular day and 1 holiday) each week during the experiment.
  3. The blood draws will be taken at approximately 11:00 am, especially prior to the first consumption of food by subjects in the TRF group. The following analyzes will be measured in plasma samples: ketones, fasting glucose, fasting insulin, hemoglobin A1c, liver function, renal function, albumin, lipid profiles, MMP-9, IL-6, TNF-alpha, exosome markers (phospho-IRS1, phospho-Tau, Abeta1-42). Metabolomic and lipidomic analyses will be performed on the baseline and 3-month time point plasma samples.
  Interventions: Behavioral: Time-restricted feeding (TRF) with dietary counseling

INTERVENTIONS:
Behavioral: Time-restricted feeding (TRF) with dietary counseling — 1. Subjects will be instructed to administer time-restricted feeding.
  2. Subjects have to compete a 3-d food record, including 2 regular day and 1 holiday. At baseline, a dietitian will provide 15 min of instruction to each participant on how to complete the food records. Subjects will be asked to measure the volume of foods consumed with household measures. The timing of food intake will be also recorded. Food records will be collected each week during the experiment and will be reviewed by the dietitian for accuracy and completeness. A database for food content will be used to calculate the total daily intake of energy, fat, protein, carbohydrate, cholesterol, and fiber. All subjects will be asked to maintain their level of physical activity throughout the entire trial.
  3. Blood withdraw will be performed prior to the first consumption of food and analyze some biochemistry data.
  Arms: Time-restricted feeding (TRF) with dietary counseling

SUMMARY:
Many preclinical studies have demonstrated the beneficial effects of intermittent fasting (IF) in a wide range of neurological and cardiovascular diseases. This pilot study aims to investigate the safety and compliance as well as efficacy of one specific IF intervention called time-restricted feeding (TRF; 16 hours fasting daily) in patients with acute ischemic stroke (AIS).

DETAILED DESCRIPTION:
Specific Aims This project is to conduct a pilot, phase II randomized clinical trial which aims to investigate the safety and compliance as well as efficacy of one specific IF intervention called time-restricted feeding (TRF; 16 hours fasting daily) in patients with acute ischemic stroke (AIS) The primary endpoint is the safety and compliance of 4 weeks of TRF in AIS patients.

The secondary endpoints are the efficacy of 4 weeks of TRF compared to normal eating (NE) on plasma and imaging biomarkers and functional outcome at 3 months post-stroke.

This study will determine whether compared to NE control:

1. TRF (16 hours fasting daily) is safe and well-tolerated in patients with AIS.
2. TRF improves functional outcome compared to NE in AIS patients. (3) TRF decreases plasma pro-inflammatory cytokines including metallopeptidase (MMP)-9, interleukin (IL)-6, and tumor necrosis factor alpha (TNF) in plasma compared to baseline and NE in AIS patients.

(4) TRF improves diffusion tensor imaging on MRI at 3 months post stroke compared to baseline and NE in AIS patients.

(5) TRF changes plasma exosome components, metabolomics and lipidomics compared to baseline and NE in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute ischemic stroke onset within 10 days
2. Age between 20-80 years.
3. Mild stroke severity (NIH stroke scale ≤ 6).

Exclusion Criteria:

1. Large hemispheric (> 1/2 middle cerebral artery territory) or cerebellar (>3 cm in diameter) infarct
2. Receiving intravenous rt-PA (alteplase) or endovascular thrombectomy
3. Severe stenosis (> 50%) or occlusion of intra/extra cranial arteries corresponding to acute ischemic stroke territory.
4. Body mass index ≤ 24.
5. Active cancer.
6. Diabetes mellitus (ex. HbA1C > 7% or taking oral hypoglycemic agent or insulin)
7. Active gastrointestinal bleeding.
8. Active infection, concurrent steroid usage or specific endocrine disorders.
9. Pre-stroke modified Rankin Scale > 2
10. Not willing to participate the trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The events of stroke in-evolution, stroke recurrence and hypoglycemia in acute ischemic stroke patients with time restricted fasting (TRF) or normal eating (NE) | 4 weeks
  1. Stroke in-evolution is defined as an increase in the NIHSS score of ≥2 points compared to initial score or the lowest score during admission, excluding other attributable medical or systemic causes.
  2. Stroke recurrence is defined as newly developed neurological deficit due to acute cerebrovascular insult during the study period.
  3. Hypoglycemia event is defined as symptomatic hypoglycemia fulfilling the criteria of Whipple's triad as symptoms known or likely to be caused by hypoglycemia, a low plasma glucose (< 60 mg/dl) measured at the time of the symptoms and relief of symptoms when the glucose is raised to normal

SECONDARY OUTCOMES:
3 months functional outcome, defined as modified Rankin Scale (mRS) <=1 as good outcome | 3 months
  Good functional outcome defined as modified Rankin Scale <=1.
Diffusion tensor imaging on MRI at baseline and 3 months post stroke | 3 months
  To evaluate the changes of diffusion tensor imaging on MRI at 3 months post stroke in TRF compared to baseline and NE in acute ischemic stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No